CLINICAL TRIAL: NCT01277705
Title: Assess Immunogenicity, Reactogenicity of GSK Biologicals'-dTpa-IPV Vaccine Versus dTpa & IPV Vaccines Administered Separately & Compared With Aventis Pasteur MSD's Td-IPV Vaccine When Administered to Healthy Adolescents & Adults
Brief Title: Comparison of GSK Biologicals' Reduced Antigen Diphtheria and Tetanus Toxoids and Acellular Pertussis- Inactivated Poliovirus Vaccine, to BoostrixTM and Inactivated Poliovirus Vaccine Administered Separately and With Revaxis®
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 711866/003
Record Dates: First submitted 2011-01-13; First posted 2011-01-17 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Tetanus; Diphtheria; Acellular Pertussis
Keywords: Booster vaccination
MeSH Terms: conditions — Tetanus; Diphtheria | interventions — Tetanus Toxoid; Boostrix

ARMS (3):
- Group A (Experimental)
  Interventions: Biological: GSK Biologicals' reduced antigen diphtheria and tetanus toxoids and acellular pertussis- inactivated poliovirus vaccine
- Group B (Experimental)
  Interventions: Biological: Boostrix™; Biological: GSK Biologicals' IPV vaccine
- Group C (Active Comparator)
  Interventions: Biological: Revaxis®

INTERVENTIONS:
Biological: GSK Biologicals' reduced antigen diphtheria and tetanus toxoids and acellular pertussis- inactivated poliovirus vaccine — Intramuscular, single
  Arms: Group A
Biological: Boostrix™ — Intramuscular, single dose
  Arms: Group B
Biological: GSK Biologicals' IPV vaccine — Intramuscular, single dose
  Arms: Group B
Biological: Revaxis® — Intramuscular, single dose
  Arms: Group C

SUMMARY:
This study will assess the immunogenicity and reactogenicity of the candidate GSK Biologicals' reduced antigen diphtheria and tetanus toxoids and acellular pertussis- inactivated poliovirus vaccine when administered to healthy subjects aged ≥ 15 years in Germany and ≥ 18 years in France compared to Boostrix™ and inactivated poliovirus vaccine administered separately, and with Revaxis®

ELIGIBILITY:
Inclusion Criteria:

* A male or female subjects aged 15 years and over (Germany), or 18 years and over (France) at the time of the vaccination.
* Written informed consent obtained.
* Free of obvious health problems Having received primary vaccination with diphtheria and tetanus vaccines to the best of his/her knowledge.
* Female subjects must not be pregnant or lactating.

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) within 30 days preceding the administration of the study vaccine dose, or planned use during the study period.
* History of previous or intercurrent diphtheria or tetanus, pertussis or polio disease in the last 10 years.
* French subjects: history of diphtheria or tetanus, pertussis or polio vaccination in the last 10 years.
* German subjects: history of diphtheria or tetanus, pertussis or polio vaccination in the last 5 years, except those subjects participating in the tetanus antibody kinetic subgroup.
* German subjects participating in the tetanus antibody kinetic subgroup: history of diphtheria or tetanus, pertussis or polio vaccination in the last 10 years.
* Administration or planned administration of a vaccine not foreseen by the study protocol during the period starting 30 days before the administration of the study vaccine dose and ending 30 days after study vaccination.
* Chronic administration or planned administration of immuno-suppressants or other immune-modifying drugs within six months or 5 half-lives (whichever is the longer) of vaccination.
* Administration of immunoglobulins and/or any blood products within the three months preceding the study vaccination or planned administration during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition,
* History of seizures or progressive neurological disease.
* Major congenital defects or serious chronic illness.
* Acute disease at the time of enrolment.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine(s).
* The following adverse experiences associated with diphtheria-tetanus-pertussis vaccination constitute absolute contraindications to further administration of diphtheria-tetanus-pertussis vaccine; if any of these adverse experiences occurred following previous vaccinations, the subject should not be included:

Absolute contraindications:

* Hypersensitivity reaction due to the vaccine.
* Encephalopathy

Precautions:

* Fever >= 40.0°C within 48 hours of vaccination not due to another identifiable cause.
* Collapse or shock-like state within 48 hours of vaccination.
* Persistent, inconsolable crying lasting >= 3 hours occurring within 48 hours of vaccination.
* Seizures with or without fever occurring within 3 days of vaccination.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 806 (Actual)
Dates: Start 2002-01; Primary Completion 2002-04 (Actual); Study Completion 2002-04 (Actual)

PRIMARY OUTCOMES:
Immunogenicity with respect to components of the study vaccines | One month after vaccination (Month 1)

SECONDARY OUTCOMES:
Immunogenicity with respect to components of the study vaccines | One month after vaccination (Month 1)
Immunogenicity with respect to some component of the study vaccines | At Day 10 after vaccination
Occurrence of solicited local and general symptoms | within 15 (Day 0-14) days after vaccination
Occurrence of unsolicited symptoms | within 30 days (Day 0-29) after vaccination
Occurrence of serious adverse events | Throughout the entire study (from Day 0 to Day 30)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Van Damme P, McIntyre P, Grimprel E, Kuriyakose S, Jacquet JM, Hardt K, Messier M, Van Der Meeren O. Immunogenicity of the reduced-antigen-content dTpa vaccine (Boostrix((R))) in adults 55 years of age and over: a sub-analysis of four trials. Vaccine. 2011 Aug 11;29(35):5932-9. doi: 10.1016/j.vaccine.2011.06.049. Epub 2011 Jun 28. PMID 21718738
- [Result] Grimprel E, von Sonnenburg F, Sanger R, Abitbol V, Wolter JM, Schuerman LM. Combined reduced-antigen-content diphtheria-tetanus-acellular pertussis and polio vaccine (dTpa-IPV) for booster vaccination of adults. Vaccine. 2005 May 25;23(28):3657-67. doi: 10.1016/j.vaccine.2005.02.013. PMID 15882526
- [Result] Wolter J et al. Boostrix polio: A new combined vaccine to fulfill emerging needs for pertussis vaccination of older age-groups. Abstract presented at the ESPID, Tampere, Finland, 26-28 May 2004.
- [Derived] Kovac M, Rathi N, Kuriyakose S, Hardt K, Schwarz TF. Immunogenicity and reactogenicity of a decennial booster dose of a combined reduced-antigen-content diphtheria-tetanus-acellular pertussis and inactivated poliovirus booster vaccine (dTpa-IPV) in healthy adults. Vaccine. 2015 May 21;33(22):2594-601. doi: 10.1016/j.vaccine.2015.03.104. Epub 2015 Apr 14. PMID 25882172
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 711866/003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 711866/003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 711866/003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 711866/003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 711866/003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 711866/003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register